CLINICAL TRIAL: NCT03405493
Title: Sleep, Wake and Light Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Kings Health Partners (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R&D2017/096
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-01

CONDITIONS: Depression; Depressive Disorder, Major; Depression, Unipolar; Depression Moderate
Keywords: Circadian Rhythm; Light Therapy; Wake Therapy; Sleep Phase Advance; Major Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder | interventions — Phototherapy; Sleep

STUDY DESIGN:
Intervention Model Description: * Both groups will receive treatment as usual.
  * Triple Chronotherapy. This consists of (a) Total Sleep Deprivation with group support on days one and two; (b) Phase Advance of Sleep over 5 days and daily Light Therapy. (c) Bright Light Therapy is given on Day 2 onwards daily.
  * Comparator Intervention: Participants will be given information on sleep hygiene and getting a good night's sleep in a written leaflet and given the opportunity to ask questions. They are then given Dim Amber Light Therapy daily for 1 week.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wake and Light Therapy (Experimental): This consists of (a) Total Sleep Deprivation with group support on days one and two; (b) Phase Advance of Sleep over 5 days and daily Light Therapy. (c) Light Therapy is given daily
  Interventions: Behavioral: Wake and Light Therapy
- Sleep and Light Therapy (Active Comparator): Participants will be given information on sleep hygiene and getting a good night's sleep. They are then given Light Therapy daily for 1 week.
  Interventions: Behavioral: Sleep and Light Therapy

INTERVENTIONS:
Behavioral: Wake and Light Therapy — Participants will be helped to change the pattern sleep by depriving participants of sleep for one night. On Day 1 participants will be supported to stay up all night and the following day at the Hospital. Participants can go to bed by 5pm at home on Day 2. Participants will need to get up by about 1am and return to the hospital to be supported to stay awake. Participants will then go to bed at 7pm on Day 3. Participants will be asked to sleep until 3am and then stay awake at home until bed at 9pm on Day 4. Participants will then get up by 5am on Day 5 and stay awake until 11pm to resume a normal sleep routine waking by 7am on Day 6. Participants will also be given a light box to use each morning. For the light box, participants will be asked to sit about one foot away from a light box. You will be free to have breakfast, read or use a computer while facing towards the light. Treatment with a light box will last 30 minutes. Participants may continue to have treatment as usual.
  Arms: Wake and Light Therapy
Behavioral: Sleep and Light Therapy — Participants will be given information and advice on how to get a good night's sleep. Participants will be also given a light box to use in the morning for 1 week. For the light box, participants will be asked to sit about one foot away from a light box. Participants will be free to have breakfast, read or use a computer while facing towards the light. Treatment with a light box will last 30 minutes when you get up. Participants may continue to have any treatment as usual (for example medication or talking therapies).
  Arms: Sleep and Light Therapy

SUMMARY:
The aim of this study is to determine if altering the pattern of one's sleep and having light therapy can speed up the treatment of depression. In the UK, the large majority of patients with depression in the NHS are treated in the community, and one of the major objectives of the study one is to determine if this therapy is a practical treatment in the community. We will be comparing two treatments:

1. Sleep Therapy and a Light Box: Participants will be given information and advice on how to get a good night's sleep. Participants will be given a light box to use in the morning for 1 week. Treatment with a light box will last 30 minutes when a person gets up. Participants may continue to have any treatment as usual (for example medication or talking therapies).
2. Wake therapy and a Light Box: Participants will be helped to change the pattern of sleep by depriving participants of sleep for one night. Participants will go bed at 5pm on the following day for 8 hours and get up at 1am. Participants' sleep will then be advanced by 2 hours each night for the next three nights. Participants will be also given a light box to use in the morning for 1 week. Treatment with a light box will last 30 minutes when participants get up. Participants may continue to have any treatment as usual (for example medication or talking therapies).

DETAILED DESCRIPTION:
* Participants will be given a wristband (Actigraph)
* Participants will be asked to complete various questionnaires and be interviewed at 1 week, 2 weeks, 4 weeks, 8 weeks and at 6 months after starting.
* Participants will be asked to make 6 extra visits to the research team at the hospital over and above those needed for normal care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Depressive Episode (ICD10 F32) or Recurrent Depressive Disorder (F33).
* Minimum score of 8 or more on the Hamilton Depression Rating Scale (6 item) (Range 0-22) (Bech,1981).
* Age 18-65
* Able to give informed consent
* Women of child bearing age may be included and no methods of contraception is required to enable inclusion into the trial.

Exclusion Criteria:

* Current diagnosis of Seasonal Affective Disorder
* Current diagnosis of anorexia nervosa or bulimia.
* Current diagnosis of an obsessive compulsive or related disorder
* Current diagnosis of post-traumatic stress disorder
* History of schizophrenia, schizoaffective disorder or bipolar disorder
* Severe cognitive impairment, dementia, intellectual disability or organic brain disorder.
* History of stimulant or hallucinogenic misuse, alcohol or substance misuse or dependence in past 3 months.
* Borderline Personality Disorder or other personality disorder considered to be the main problem.
* Duration of depression more than 2 years.
* Significant risk of suicide that requires hospitalisation.
* Severe eye disease or cataracts or traumatic injury or visual impairment affecting both eyes.
* History of epilepsy, uncontrolled severe headaches, or stroke as this may lower seizure threshold through sleep deprivation.
* Unstable medical condition that would make wake therapy intolerable
* Untreated sleep disorder such as obstructive sleep apnoea or narcolepsy
* Use of photo-sensitizing drugs.
* Current night-shift work.
* Non-English speaker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited per month/Adherence to the protocol | Week 1
  To compare the rate of recruitment and adherence to the treatments in both groups

SECONDARY OUTCOMES:
MINI International Neuropsychiatric Interview Version 5.0 | Baseline
  To determine diagnosis by DSM-IV criteria
Hamilton Depression Rating Scale | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  To compare the effects on observer rated depressive symptoms in both groups
Clinical Global Impression and Improvement Scale (Guy, 1976) | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  To compare the effects on observer rated clinical impression in both groups
Quick Inventory of Depressive Symptomatology -SR Version (Triveni et al., 2004) Questionnaire | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  To compare the effects on subjective depressive symptoms in both groups
Brief Ruminative Response Scale (Topper et al, 2014). Questionnaire | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  To compare the effects on measures of subjective rumination in both groups
Pittsburgh Sleep Index (Bysse et al., 1999) Questionnaire | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  To compare the effects on subjective sleep quality in both groups
Euroquol 5D (1990) Questionnaire | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  To compare the effects on subjective general quality of life in both groups
To check the amount of current antidepressant use | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  Amount of antidepressant drugs (in mg of antidepressant equivalents) (Hayasaka et al., 2015) or benzodiazepine drugs (in mg of diazepam equivalents)
To check the amount of current psychotherapy use | Baseline, and at 1, 2, 4, 8 weeks and 6-month post-randomisation
  The amount of Cognitive Behaviour Therapy or any other counselling or psychotherapy (number of hours)
Daily sleep diary | 3 days pre-randomisation and 7 days post-randomisation
  A subjective measure of total sleep time
Credibility and Expectancy Questionnaire (Devilly, 2000). | Baseline
  A measure of the credibility of the intervention
Morning/Evening Questionnaire | 3 days pre-randomisation
  A measure of morning/evening preference
Wrist actigraph from GeneActiv daily (Physiological parameter) | 3 days pre-randomisation and 7 days post-randomisation.
  A measure of the sleep/wake activity, which correlates with the gold standard of sleep physiology (polysomnography).

CONTACTS AND LOCATIONS:
Overall Officials: David Veale, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03405493/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03405493/ICF_001.pdf